CLINICAL TRIAL: NCT03268824
Title: Impact of Epileptic Discharge on the Structural Connectivity of the Developing Brain: Combination of Intracerebral Stereotactic Electroencephalography Recording and Diffusion Tensor Imaging in Children With Drug-resistant Focal Epilepsy
Brief Title: Impact of Epileptic Discharge on the Structural Connectivity of the Developing Brain
Acronym: EPITRACT
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: VDR_2017_1
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Epilepsies, Focal; Pediatrics; Drug Resistant Epilepsy
MeSH Terms: conditions — Epilepsies, Partial; Drug Resistant Epilepsy | interventions — Electroencephalography; Diffusion Tensor Imaging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children / adolescents with drug-resistant focal epilepsy
  Interventions: Device: Electroencephalogram (EEG); Device: Diffusion Tensor imaging; Other: Language assessment
- Children / adolescents without drug-resistant focal epilepsy
  Interventions: Device: Diffusion Tensor imaging; Other: Language assessment

INTERVENTIONS:
Device: Electroencephalogram (EEG) — Intracerebral electroencephalogram (EEG) will be analysed to quantify the intensity of epileptic discharge (the epileptogenicity index) on each electrode contact (only for children with focal epilepsy).
  Groups: Children / adolescents with drug-resistant focal epilepsy
Device: Diffusion Tensor imaging — We will perform Diffusion Tensor imaging in order to relate tractography measures to seizure recordings. Loss of connectivity (or disconnections) will be determined with diffusion tractography for each brain region. Then we will correlate the degree of epileptogenicity with the number of disconnections.
Other: Language assessment — The language assessment will be adapted to the age of the child, with a predominant neuropsychological component.

SUMMARY:
Focal epilepsy is associated with widespread alterations in structural brain connectivity, often present at the disease onset and related to learning disabilities. Whether ongoing seizure activity contributes to network pathology is a matter of debate. This study intends to measure the impact of seizures on structural connectivity on a local and on a global level. In children examined with intracerebral electrodes to evaluate whether a surgical cure can be proposed, we combine intracerebral stereotactic electroencephalography (EEG) recordings with diffusion weighted imaging of white matter fibers. On the local level, the study will quantify the number of deficient connections in the seizure onset zone. On a global level, the study will compare the white matter fibers of the left and right hemisphere to probe whether physiological language lateralization is preserved.

DETAILED DESCRIPTION:
Drug-resistant focal epilepsy is a debilitating disease as it is often accompanied by learning disabilities and behavioral disorders, that can be present at the disease onset and have ample repercussions on the child's quality of life.

Despite a focal onset of seizures, the dysfunction of the cerebral networks is diffuse. Structural brain connectivity can be measured with diffusion tractography, which has shown evidence of widespread network pathology in focal epilepsy, probably explaining the associated learning disabilities. Whether ongoing seizure activity further modifies network wiring and possibly generates abnormal pathways along the routes of seizure propagation is a matter of debate.

The study intends to probe the effect of seizures on cerebral connectivity, both on a local and on a global level. Children who undergo presurgical evaluation to probe whether their epilepsy can be cured by surgery are recorded with implanted intracerebral electrodes for clinical purposes. A diffusion Magnetic Resonance Imaging will be performed prior to implantation in order to relate tractography measures to seizure recordings. On the local level, intracerebral electroencephalogram (EEG) will be analysed to quantify the intensity of epileptic discharge (the epileptogenicity index) on each electrode contact. Loss of connectivity (or disconnections) is determined with diffusion tractography for each brain region. Then correlation between the degree of epileptogenicity and with the number of disconnections will be studied.

On a global level, the study will quantify all white matter fibers within the language area (Broca's) in the left and the corresponding area in the right hemisphere. The difference between hemispheres yields us the lateralization index. The secondary outcome probes whether children with focal epilepsy have atypical language organization, as a measure of diffuse changes in brain wiring.

ELIGIBILITY:
Inclusion Criteria:

- Drug resistant focal epilepsy

Inclusion Criteria for control patients:

- without drug resistant focal epilepsy

Exclusion Criteria:

* Severe mental retardation (IQ < 50)
* Lack of French-language skills
* Contraindications to MRI
* Bi-hemispherical epilepsy or affecting multiple lobes

Exclusion Criteria for control patients:

* Severe mental retardation (IQ < 50)
* Lack of French-language skills
* Contraindications to MRI
* Congenital pathology altering cerebral connectivity
* Parenchymal brain lesions
* Unilateral or bilateral blindness
* Unilateral or bilateral deafness
* Autistic disorders

Ages: 18 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children/adolescents with drug resistant focal epilepsy.
Sampling Method: Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2017-12-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Correlation between the number of cerebral disconnections and the epileptogenicity index | Baseline
  The epileptogenicity index is based on measurement of the intensity of rapid frequency discharges in relation to the cerebral activity outside the seizures.

CONTACTS AND LOCATIONS:
Overall Officials: Vera Dinkelacker, MD PhD, Principal Investigator — Fondation Ophtalmologique A. de Rothschild
Locations (1):
- Fondation Ophtalmologique A. de Rothschild, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided